CLINICAL TRIAL: NCT03280979
Title: Comparison Between Rescue Regimen and High Dose Methotrexate in the Managment of Presistent Gestational Trophoplastic Neoplasia :( A Randomized Controlled Trial )
Brief Title: Rescue Regimen and High Dose Methotrexate in Management of Presistent Gestational Trophoplastic Neoplasia
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Zahraa Magdy, principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RR&HDMPGTN
Record Dates: First submitted 2017-09-11; First posted 2017-09-13 (Actual); Last update posted 2017-09-13 (Actual); Status verified 2017-09

CONDITIONS: Gestational Trophoblastic Disease
MeSH Terms: conditions — Gestational Trophoblastic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group1 (Experimental): In the rescue regimen , we administer MTX in an eight-day treatment regimen consisting of four administrations of MTX given at 1 mg/kg I.M. every other day with folinic acid 0.1 mg/kg I.M,. given on intervening days.
  Interventions: Drug: rescue regimen
- study group2 (Experimental): In the high dose MTX protocol, the patients will receive 100 mg/m2 intravenous (IV) MTX bolus followed by 200 mg/m2IV MTX infused over 12 hours followed by folinic acid
  Interventions: Drug: high dose methotrxate

INTERVENTIONS:
Drug: rescue regimen — In the rescue regimen , we administer MTX in an eight-day treatment regimen consisting of four administrations of TX given at 1 mg/kg I.M. every other day with folinic acid 0.1 mg/kg I.M,. given on intervening days.
  Arms: study group1
Drug: high dose methotrxate — In the high dose MTX protocol, the patients will receive 100 mg/m2 intravenous (IV) MTX bolus followed by 200 mg/m2IV MTX infused over 12 hours followed by folinic acid
  Arms: study group2

SUMMARY:
Gestational trophoblastic neoplasia (GTN) are malignant lesions that arise from abnormal proliferation of placental trophoblast. The pathologic conditions that make up this entity include invasive partial and complete hydatidiform mole, choriocarcinoma, placental site trophoblastic tumor (PSTT), and epithelioid trophoblastic tumor (ETT). GTN often arises after molar pregnancies but can also occur after any gestation including miscarriages and term pregnancies. In the United States, hydatidiform moles are observed in approximately 1/600 therapeutic abortions and 1/1000-2000 pregnancies . Most cases of GTN are diagnosed when the serum hCG levels plateau or rise in patients being observed after the diagnosis of hydatidiform mole.These malignancies are highly susceptible to chemotherapy and it is often possible to achieve cure while preserving the woman's reproductive function

DETAILED DESCRIPTION:
When reporting GTN data, it is useful to use both the FIGO anatomic staging system and prognostic scoring system . A FIGO score of 6 or less indicates low-risk GTN whereas a score of 7 or more identifies high-risk disease.

Table 1- FIGO Anatomical staging of gestational trophoblastic neoplasia:

Stage I Disease confined to the uterus Stage II Disease extends to the outside of the uterus, but is limited to the genital structures Stage III Disease extends to the lungs, with or without genital tract involvement Stage IV All other metastatic sites

Table 2- FIGO Scoring system:

FIGO SCORING 0 1 2 4 Age (years) Antecedent pregnancy Interval months from end of index pregnancy to treatment Pretreatment serum hCG (iu/l) Largest tumour size, including uterus Site of metastases Number of metastases Previous failed chemotherapy <40 ≥40 - - mole abortion term <4 4-6 7-12 >12 <1000 1000-10000 10000-100000 >100000 <3cm 3-4cm ≥5 - Lung spleen&kidney GIT liver&brain

* 1-4 5-8 >8
* - 1 drug 2 or more drugs

RCOG guidelines (No. 38February 2010 ) recommends the use of rescue regimen of alternating methotrexate( MTX) and leucoverin for 8 days (class D). However, several protocols using MTX were described. No prospective randomised controlled trials have been done to compare the efficacy of resue regimen with the ther protocols. In a retrospective study done showed that high dose methotrexate regimen is more effective than the rescue regimen.

In addition, several concerns have been raised towards the use of leucoverin with methotrexate, although reducing the side effects, however, it may increase the resistence to the effect of MTX .

On the other hand, High dose regimen offers a less hospital stay which may be more convenient to the patients, together with the same incidence of side effects.

In our study we are going to compare the efficacy and tolerance of both regimens in patients diagnosed to have low risk PGTN.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-50
* BW: 50-100 kg
* willing and consenting to be enrolled in the study
* Absence of active vaginal bleeding which requires surgical intervention • - WHO score <6

Exclusion Criteria:

* Renal and liver dysfunction or blood dyscariasis
* high risk persistent gestational trophoblastic disease.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 170 (Estimated)
Dates: Start 2017-10 (Estimated); Primary Completion 2019-07 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
cure rate | 12 month
  cure rate till B hcG is negative and then 2 consolidation regimens

SECONDARY OUTCOMES:
decline in Bhcg | 12 month
  Number of cycles for decline in BhCG

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol